CLINICAL TRIAL: NCT01223742
Title: ORAL ACETYL-L-CARNITINE THERAPY REDUCES FATIGUE IN HEPATIC ENCEPHALOPATHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Other Study IDs: 8-12-00 B
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2000-12

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACETYL-L-CARNITINE (Experimental)
  Interventions: Dietary Supplement: ACETYL-L-CARNITINE
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: ACETYL-L-CARNITINE — 2 g acetylcarnitine taken orally twice a day.
  Arms: ACETYL-L-CARNITINE
Drug: placebo — placebo twice per day
  Arms: placebo

SUMMARY:
The aim of this study was to evaluate the effect of exogenous ALC on the both physical and mental fatigue in mild and moderate encephalopatic patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Chronic hepatitis with spontaneous manifest HE (mental state grade 1 or 2 according to the West Haven criteria) and an NCT-A performance time >30 seconds;
* 2) Hyperammonemia (venous ammonia concentration >50 mmol/L);
* 3) Cooperative, hospitalised, adult patients with liver cirrhosis diagnosed by clinical, histological and ultrasonographic findings (reduced dimensions of the liver as well as splenomegaly) and oesophageal varices at stage II and III observed by endoscopy.

Exclusion Criteria:

* 1) Major complications of portal hypertension, such as gastrointestinal blood loss, hepatorenal syndrome or bacterial peritonitis;
* 2) Acute superimposed liver injury;
* 3) Patient with other neurological disease and metabolic disorders, diabetes mellitus, unbalanced heart failure and/or respiratory failure or end-stage renal disease;
* 4) Alcoholic -toxic cirrhosis because toxic brain damage may interfere with the assessment of HE;
* 5) Severe HE;
* 6) Administration of anti-HE medications such as neomycin, branched-chain amino acids;
* 7) Any additional precipitating factors such as high protein intake (additional high-protein meals), constipation or intake of psycho stimulants, sedatives, antidepressants, benzodiazepines, or benzodiazepines-antagonists (flumazenil), beta-adrenergic blockers, neuromuscular blocking agents, certain antibiotics;
* 8) Patients with fever, sepsis or shock were also excluded to avoid variations caused by body temperature;
* 9) Illiteracy.

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Locations (1):
- Cannizzaro Hospital, Catania, Italy

REFERENCES:
- [Derived] Malaguarnera M, Vacante M, Giordano M, Pennisi G, Bella R, Rampello L, Malaguarnera M, Li Volti G, Galvano F. Oral acetyl-L-carnitine therapy reduces fatigue in overt hepatic encephalopathy: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2011 Apr;93(4):799-808. doi: 10.3945/ajcn.110.007393. Epub 2011 Feb 10. PMID 21310833